CLINICAL TRIAL: NCT05160441
Title: A Prospective, Single-blind, Randomized, Multi-Center Study Comparing Platelet Rich Plasma and Corticosteroid for Patients With Glenohumeral Osteoarthritis in the Military and Civilian Population
Brief Title: Comparing Platelet Rich Plasma and Corticosteroid for Military & Civilian Patients With Glenohumeral Osteoarthritis
Acronym: PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sean Slaven, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WRNMMC-2021-0345
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis of the Shoulder; Corticosteroid; PRP; Pain
MeSH Terms: conditions — Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Platelet Rich Plasma Injection Group (Experimental): Minimum 2cc Leukocyte Poor Platelet Rich Plasma
  Interventions: Biological: Platelet Rich Plasma Injection
- Corticosteroid Injection Group (Active Comparator): 5cc Normal Saline + 2cc 10 mg/ml Triamcinolone Acetonide (Kenalog)
  Interventions: Biological: Corticosteroid Injection
- Delayed Platelet Rich Plasma Injection Group upon Corticosteroid Injection Failure (Experimental): If a participant does not have any benefit from the corticosteroid injection by the six-week follow-up time point, then that participant will be eligible for a platelet rich plasma injection.
  Interventions: Biological: Delayed Platelet Rich Plasma Injection After Corticosteroid Injection Failure

INTERVENTIONS:
Biological: Platelet Rich Plasma Injection — Minimum 2cc Leukocyte Poor Platelet Rich Plasma
  The PRP will be prepared by drawing 60cc blood from the participant through venipuncture, spinning the blood sample in a centrifuge and then injecting the platelet rich plasma (approximately 2-5cc or max collected) into the study shoulder using ultrasound guidance. This sample will be prepared by the study provider (physician assistant or physician). Any leftover blood will be safely discarded per standard protocols.
  Arms: Platelet Rich Plasma Injection Group
Biological: Corticosteroid Injection — 5cc Normal Saline + 2cc 10 mg/ml Triamcinolone Acetonide (Kenalog)
  Arms: Corticosteroid Injection Group
Biological: Delayed Platelet Rich Plasma Injection After Corticosteroid Injection Failure — Participants randomized to the corticosteroid injection (CSI) group who report no improvement in their pain level at the 6 week post-CSI visit will be unblinded to their study injection (CSI) and will be offered the option to stay in the study and receive Platelet Rich Plasma injection.
  Arms: Delayed Platelet Rich Plasma Injection Group upon Corticosteroid Injection Failure

SUMMARY:
Shoulder arthroplasty provides successful improvement in pain and function for the treatment of end stage osteoarthritis (OA) of the shoulder in the older patient population (Sanchez 2008, Sampson 2010, Kon 2012, Fitzpatrick 2017). However, the optimal non-operative treatment for shoulder OA in the young active duty and civilian populations has yet to be determined. Although corticosteroid injections (CSI) are a viable option with diagnostic and short-term therapeutic benefit in glenohumeral OA, steroid does little to address the underlying pathology and confers risk of adjacent tendon failure (Kon 2009, Gosens 2011, Monto 2014, Tietze 2014). Platelet-rich plasma (PRP) derived from autologous blood, however, has the potential to enhance soft tissue healing as previously observed in muscles and tendons (Sanchez 2005, Randelli 2008, Hall 2009). PRP contains growth factors purported to safely facilitate local tissue regeneration as corroborated in multiple clinical studies investigating tendinopathy (Virchenko 2006, Kesikburun 2013, Fitzpatrick 2017, Schwitzguebel 2019). PRP is a promising concept to bridge the gap between conventional non-operative measures and surgical arthroscopy or arthroplasty options in a high functioning patient population with refractory disease. However, clinical literature elucidating the effects of intra-articular leukocyte-poor PRP (LP-PRP) injections in large joint degenerative OA has been slower to emerge, lacking substantiated data due to small sample sizes and treatment variability. Therefore, high level evidence-based studies remain critical in ascertaining the therapeutic value and clinical efficacy of LP-PRP in glenohumeral OA in order to establish standard of care protocols and guide systematic implementation.

DETAILED DESCRIPTION:
Shoulder arthroplasty provides successful improvement in pain and function for the treatment of end stage osteoarthritis (OA) of the shoulder in the older patient population (Sanchez 2008, Sampson 2010, Kon 2012, Fitzpatrick 2017). However, the optimal non-operative treatment for shoulder OA in the young active duty and civilian populations has yet to be determined. Although corticosteroid injections (CSI) are a viable option with diagnostic and short-term therapeutic benefit in glenohumeral OA, steroid does little to address the underlying pathology and confers risk of adjacent tendon failure (Kon 2009, Gosens 2011, Monto 2014, Tietze 2014). Platelet-rich plasma (PRP) derived from autologous blood, however, has the potential to enhance soft tissue healing as previously observed in muscles and tendons (Sanchez 2005, Randelli 2008, Hall 2009). PRP contains growth factors purported to safely facilitate local tissue regeneration as corroborated in multiple clinical studies investigating tendinopathy (Virchenko 2006, Kesikburun 2013, Fitzpatrick 2017, Schwitzguebel 2019). PRP is a promising concept to bridge the gap between conventional non-operative measures and surgical arthroscopy or arthroplasty options in a high functioning patient population with refractory disease. However, clinical literature elucidating the effects of intra-articular leukocyte-poor PRP (LP-PRP) injections in large joint degenerative OA has been slower to emerge, lacking substantiated data due to small sample sizes and treatment variability. Therefore, high level evidence-based studies remain critical in ascertaining the therapeutic value and clinical efficacy of LP-PRP in glenohumeral OA in order to establish standard of care protocols and guide systematic implementation.

Although commonly used corticosteroid injections have shown some clinical benefit, there are known deleterious effects from steroid use, which include accelerated osteoarthritis progression, cartilage toxicity, and increased risk of septic arthritis. In addition to this, multiple studies demonstrate corticosteroids confers risk of adjacent tendon failure (Kon 2009, Gosens 2011, Monto 2014, Tietze 2014). There is also a concern that multiple corticosteroid injections increase the risk of fat atrophy, skin pigment changes, and tissue thinning if placed incorrectly in the more superficial tissue of the shoulder. These negative findings associated with corticosteroid injections have prompted ongoing research into alternative orthobiologic treatments that provide short to medium duration benefit for patients with osteoarthritis.

Conversely, Leukocyte-Poor Platelet-Rich Plasma (LP-PRP), derived from autologous blood, has demonstrated safety and efficacy in multiple pre-clinical, randomized controlled clinical trials, and meta-analysis studies in the other large joints, causing slow acceptance in the medical community to utilize this as a treatment option, despite its increased cost compared to corticosteroid injection (Campbell 2015, Cavallo 2014, Lai 2015, Laudy 2015, Patel 2013, Smith 2016, Tietze 2014, Piuzzi 2019). However, clinical literature elucidating the effects of intraarticular leukocyte-poor PRP (LP-PRP) injections in shoulder joint degenerative OA has been slower to emerge, lacking substantiated data due to small sample sizes and treatment variability. Therefore, high level evidence-based studies remain critical in ascertaining the therapeutic value and clinical efficacy of LP-PRP in glenohumeral OA in order to establish standard of care protocols and guide systematic implementation. PRP is a promising concept to bridge the gap between conventional non-operative measures and surgical arthroscopy or arthroplasty options in a high functioning patient population with refractory disease.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible
* Male or female, aged 18 to 70 years (inclusive)
* Presenting symptoms of shoulder pain caused by mild to moderate Shoulder OA as defined by Samilson Prieto criteria on a standard anterior-posterior (AP) Xray series
* BMI < 40
* Willing and able to give voluntary informed consent to participate in this investigation
* Glenohumeral joint osteoarthritis that has been refractory to standard care treatments

Exclusion Criteria:

* Patients who have received shoulder intraarticular or subacromial injection(s) in the last 3 months
* Patients who have undergone arthroscopic surgery on the study shoulder within the past year
* Patients who have undergone arthroplasty on the study shoulder
* Diabetes (Type 1 or II)
* Inflammatory arthropathies
* Fibromyalgia or chronic fatigue syndrome
* Female patient who is pregnant or nursing
* Patients taking narcotics
* Patients with planned deployment or separation from the military within 12 months
* Any other serious medical condition(s) that might preclude optimal outcome and/or interfere with participation such as intra-articular sepsis, bacteremia, fracture, joint instability, rheumatoid arthritis, osteoporosis, cancer, and coagulopathy
* Patients who have had an adverse reaction to a previous corticosteroid or PRP injection either documented in the medical record or shared by the patient during screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Change in the Single Assessment Numeric Evaluation (SANE) from before injection to after injection | Pre-injection (baseline) and then post-injection at 3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The SANE score is a validated patient reported outcome measure. It is a single question score that asks, "how would you rate your condition today as a percentage of normal (0% to 100% scale with 100% being normal)?" The SANE score is collected as standard of care.
Change in the American Shoulder and Elbow Surgeons Standardized Shoulder Form (ASES) from before injection to after injection | Pre-injection (baseline) and then post-injection at 3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points
Change in the Visual Analogue Scale (VAS) from before injection to after injection | Pre-injection (baseline) and then post-injection at 3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Change in the Veterans RAND 12-Item Health Survey (VR-12) from before injection to after injection | Pre-injection (baseline) and then post-injection at 3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The VR-12 comprises 12 questions that correspond to eight domains of health, including general health perceptions, physical functioning, role limitations because of physical problems, role limitations because of emotional problems, bodily pain, vitality, social functioning, and mental health.
Change in the Western Ontario Osteoarthritis Shoulder Index (WOOS) from before injection to after injection | Pre-injection (baseline) and then post-injection at 3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The WOOS is a patient-administrated, disease-specific questionnaire for measurement of the quality-of-life of patients with osteoarthritis.7 It provides scores on four domains: (1) physical symptoms; (2) sport, recreation, and work; (3) lifestyle; and (4) emotions. Each question is answered using a visual analog scale with a possible score ranging from 0 to 100. There are 19 questions, and the total score ranges from 0 to 1900. A score of 1900 signifies that the patient has an extreme decrease in the shoulder-related quality of life, whereas a score of 0 signifies that the patient has no decrease in shoulder-related quality of life.
Change in range of motion (ROM) from before injection to after injection | Pre-injection (baseline) and then post-injection at 6 weeks, 3 months, 6 months, 12 months, and 24 months
  Testing the range of motion (ROM) of the shoulder in different directions. If movement in a specific direction is painful or limited, this may signify that pathology is present in a specific structure of the shoulder. Common ROM tests include: forward flexion, abduction, cross-body adduction, external rotation, extension, internal rotation, scapular motion

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be shared with anyone. Only aggregate results will be shared publicly.

REFERENCES:
- [Background] Centeno CJ, Al-Sayegh H, Bashir J, Goodyear S, Freeman MD. A prospective multi-site registry study of a specific protocol of autologous bone marrow concentrate for the treatment of shoulder rotator cuff tears and osteoarthritis. J Pain Res. 2015 Jun 5;8:269-76. doi: 10.2147/JPR.S80872. eCollection 2015. PMID 26089699
- [Background] Fitzpatrick J, Bulsara M, Zheng MH. The Effectiveness of Platelet-Rich Plasma in the Treatment of Tendinopathy: A Meta-analysis of Randomized Controlled Clinical Trials. Am J Sports Med. 2017 Jan;45(1):226-233. doi: 10.1177/0363546516643716. Epub 2016 Jul 21. PMID 27268111
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Background] Hak A, Rajaratnam K, Ayeni OR, Moro J, Peterson D, Sprague S, Bhandari M. A Double-Blinded Placebo Randomized Controlled Trial Evaluating Short-term Efficacy of Platelet-Rich Plasma in Reducing Postoperative Pain After Arthroscopic Rotator Cuff Repair: A Pilot Study. Sports Health. 2015 Jan;7(1):58-66. doi: 10.1177/1941738114548413. PMID 25553214
- [Background] Hall MP, Band PA, Meislin RJ, Jazrawi LM, Cardone DA. Platelet-rich plasma: current concepts and application in sports medicine. J Am Acad Orthop Surg. 2009 Oct;17(10):602-8. doi: 10.5435/00124635-200910000-00002. PMID 19794217
- [Background] Kesikburun S, Tan AK, Yilmaz B, Yasar E, Yazicioglu K. Platelet-rich plasma injections in the treatment of chronic rotator cuff tendinopathy: a randomized controlled trial with 1-year follow-up. Am J Sports Med. 2013 Nov;41(11):2609-16. doi: 10.1177/0363546513496542. Epub 2013 Jul 26. PMID 23893418
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Kon E, Filardo G, Drobnic M, Madry H, Jelic M, van Dijk N, Della Villa S. Non-surgical management of early knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2012 Mar;20(3):436-49. doi: 10.1007/s00167-011-1713-8. Epub 2011 Oct 25. PMID 22037809
- [Background] Randelli PS, Arrigoni P, Cabitza P, Volpi P, Maffulli N. Autologous platelet rich plasma for arthroscopic rotator cuff repair. A pilot study. Disabil Rehabil. 2008;30(20-22):1584-9. doi: 10.1080/09638280801906081. PMID 18608363
- [Background] Monto RR. Platelet-rich plasma efficacy versus corticosteroid injection treatment for chronic severe plantar fasciitis. Foot Ankle Int. 2014 Apr;35(4):313-8. doi: 10.1177/1071100713519778. Epub 2014 Jan 13. PMID 24419823
- [Background] Sampson S, Reed M, Silvers H, Meng M, Mandelbaum B. Injection of platelet-rich plasma in patients with primary and secondary knee osteoarthritis: a pilot study. Am J Phys Med Rehabil. 2010 Dec;89(12):961-9. doi: 10.1097/PHM.0b013e3181fc7edf. PMID 21403592
- [Background] Sanchez, M., Anitua, E., & Andia, I. (2005, May). Application of autologous growth factors on skeletal muscle healing. In 2nd World Congress on Regenerative Medicine. Podium Presentation.
- [Background] Sanchez M, Anitua E, Orive G, Mujika I, Andia I. Platelet-rich therapies in the treatment of orthopaedic sport injuries. Sports Med. 2009;39(5):345-54. doi: 10.2165/00007256-200939050-00002. PMID 19402740
- [Background] Schwitzguebel AJ, Kolo FC, Tirefort J, Kourhani A, Nowak A, Gremeaux V, Saffarini M, Ladermann A. Efficacy of Platelet-Rich Plasma for the Treatment of Interstitial Supraspinatus Tears: A Double-Blinded, Randomized Controlled Trial. Am J Sports Med. 2019 Jul;47(8):1885-1892. doi: 10.1177/0363546519851097. Epub 2019 Jun 4. PMID 31161947
- [Background] Sanchez M, Anitua E, Azofra J, Aguirre JJ, Andia I. Intra-articular injection of an autologous preparation rich in growth factors for the treatment of knee OA: a retrospective cohort study. Clin Exp Rheumatol. 2008 Sep-Oct;26(5):910-3. PMID 19032827
- [Background] Tietze DC, Geissler K, Borchers J. The effects of platelet-rich plasma in the treatment of large-joint osteoarthritis: a systematic review. Phys Sportsmed. 2014 May;42(2):27-37. doi: 10.3810/psm.2014.05.2055. PMID 24875970
- [Background] Virchenko O, Aspenberg P. How can one platelet injection after tendon injury lead to a stronger tendon after 4 weeks? Interplay between early regeneration and mechanical stimulation. Acta Orthop. 2006 Oct;77(5):806-12. doi: 10.1080/17453670610013033. PMID 17068715
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT05160441/ICF_001.pdf